CLINICAL TRIAL: NCT00706654
Title: A 38-week, Multicenter, Randomized, Double-blind, Active-controlled Study to Evaluate the Efficacy, Safety, and Tolerability of an Intramuscular Depot Formulation of Aripiprazole (OPC-14597) as Maintenance Treatment in Patients With Schizophrenia
Brief Title: Intramuscular Depot Formulation of Aripiprazole as Maintenance Treatment in Patients With Schizophrenia
Acronym: ASPIRE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 31-07-247
Record Dates: First submitted 2008-06-25; First posted 2008-06-27 (Estimated); Results first posted 2013-08-14 (Estimated); Last update posted 2013-08-14 (Estimated); Status verified 2013-07

CONDITIONS: Schizophrenia
Keywords: Aripiprazole; Intramuscular (IM) depot; Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Aripiprazole depot 300 or 400 mg (Experimental): Patients received aripiprazole 300 mg or 400 mg depot intramuscularly every 28 days for 38 weeks.
  Interventions: Drug: Aripiprazole depot 300 or 400 mg; Drug: Placebo tablets
- Aripiprazole 10-30 mg orally (Active Comparator): Patients received aripiprazole 10-30 mg orally daily for 38 weeks.
  Interventions: Drug: Aripiprazole 10-30 mg orally; Drug: Placebo depot
- Aripiprazole depot 25 or 50 mg (Experimental): Patients received aripiprazole 25 mg or 50 mg depot intramuscularly every 28 days for 38 weeks.
  Interventions: Drug: Aripiprazole depot 25 or 50 mg; Drug: Placebo tablets

INTERVENTIONS:
Drug: Aripiprazole depot 300 or 400 mg — Aripiprazole depot was supplied in 400 mg lyophilized vials. Patients received aripiprazole 300 mg if they were unable to tolerate aripiprazole 400 mg.
  Other Names: Abilify
  Arms: Aripiprazole depot 300 or 400 mg
Drug: Aripiprazole 10-30 mg orally — Aripiprazole was supplied as 10, 15, and 20 mg tablets. The dose that the patient received was based on the investigator's judgment and the subject's clinical need.
  Other Names: Abilify
  Arms: Aripiprazole 10-30 mg orally
Drug: Aripiprazole depot 25 or 50 mg — Aripiprazole depot was supplied in 200 mg lyophilized vials. Patients received aripiprazole 25 mg if they were unable to tolerate aripiprazole 50 mg.
  Other Names: Abilify
  Arms: Aripiprazole depot 25 or 50 mg
Drug: Placebo depot — Placebo depot was supplied in lyophilized vials.
  Arms: Aripiprazole 10-30 mg orally
Drug: Placebo tablets — Placebo tablets were identical in appearance to the aripiprazole tablets.
  Arms: Aripiprazole depot 25 or 50 mg; Aripiprazole depot 300 or 400 mg

SUMMARY:
The purpose of the this trial is to evaluate the efficacy, safety, and tolerability of an intramuscular (IM) depot formulation of aripiprazole as maintenance treatment in patients with schizophrenia

The trial is designed into three treatment phases. Phase 1 is designed to allow for a subject to be converted from the current anti-psychotic treatment to oral non-generic aripiprazole monotherapy (oral conversion phase from 4 to 6 weeks). During Phase 2 the subject will be stabilized on oral non-generic aripiprazole monotherapy. Once the subject is stabilized in Phase 2 (oral stabilization phase from minimum 8 weeks to maximum 28 weeks), they are eligible to be randomized into the double-blind IM depot maintenance phase, Phase 3. During Phase 3, the subject will be assessed for exacerbation of psychotic symptoms and impending relapse for up to 38 weeks.

DETAILED DESCRIPTION:
This will be a randomized, double-blind, active-controlled study consisting of a screening phase and 3 treatment phases. Eligibility will be determined during a screening phase of 2 to 42 days. Subjects currently receiving oral treatment with an anti-psychotic other than non-generic aripiprazole will enter Phase 1, and subjects with a lapse in aripiprazole or other anti-psychotic treatment at the time of study entry ("lapse" defined as > 3 consecutive days without medication) will enter directly into Phase 2.

During Phase 1 (oral conversion), subjects will be cross-titrated during weekly visits from other anti-psychotics to oral non-generic aripiprazole monotherapy over a minimum of 4 weeks and a maximum of 6 weeks. During Phase 2 (that will be a minimum of 8 weeks and a maximum of 28 weeks in duration), subjects will be assessed bi-weekly and stabilized on an oral dose of aripiprazole ranging from 10 mg to 30 mg daily. After stability criteria are met at Phase 2, subjects are eligible to be randomized into the double-blind IM depot maintenance phase, Phase 3. Subjects will be randomized with a 2:2:1 (aripiprazole IM depot 300-400 mg monthly, oral aripiprazole 10-30 mg daily, aripiprazole IM depot 25-50 mg monthly). During Phase 3 subjects will be assessed for impending relapse/exacerbation of psychotic symptoms. If a subject is identified with impending relapse/exacerbation of psychotic symptoms, they will be withdrawn from the trial and given the opportunity to enroll into an open-label aripiprazole IM depot trial, 31-08-248 (NCT00731549). Alternatively, any subject that discontinues in Phase 3 (up to and including Week 38) will have the option to enroll into an open-label aripiprazole IM depot trial, 31-08-248 (NCT00731549).

The enrollment figure includes re-screened patients.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are able to provide written informed consent and/or consent obtained from a legally acceptable representative (as required by Institutional Review Board/Independent Ethics Committee [IRB/IEC]), prior to the initiation of any protocol-required procedures.
* Male and female subjects 18 to 60 years of age, inclusive, at time of informed consent.
* Subjects with a current diagnosis of schizophrenia as defined by Diagnostic and Statistical Manual of Mental Disorders, version 4, Text Revision (DSM-IV-TR) criteria and a history of the illness for at least 3 years prior to screening.
* Subjects who, in the investigator's judgment, require chronic treatment with an anti-psychotic medication.
* Subjects able to understand the nature of the study and follow protocol requirements, including the prescribed dosage regimens, tablet ingestion, IM depot injection, discontinuation of prohibited concomitant medications, who can read and understand the written word in order to complete patient-reported outcome measures, and who can be reliably rated on assessment scales.

Exclusion Criteria:

* Subjects with a current DSM-IV-TR diagnosis other than schizophrenia, including schizoaffective disorder, major depressive disorder, bipolar disorder, delirium, dementia, amnestic, or other cognitive disorders. Also, subjects with borderline, paranoid, histrionic, schizotypal, schizoid, or antisocial personality disorder.
* Subjects with schizophrenia that are considered resistant/refractory to antipsychotic treatment by history or response only to clozapine.
* Subjects with a significant risk of violent behavior or a significant risk of committing suicide based on history or investigator's judgment.
* Subjects who currently meet DSM-IV-TR criteria for substance dependence; including alcohol and benzodiazepines, but excluding caffeine and nicotine, or 2 positive drug screens for cocaine.
* Subjects who are known to be allergic, intolerant, or unresponsive to prior treatment with aripiprazole or other quinolinones, or hypersensitivity to anti-psychotic agents, including aripiprazole.
* Subjects with a history of neuroleptic malignant syndrome or clinically significant tardive dyskinesia at screening.
* Subjects with uncontrolled thyroid function abnormalities.
* Subjects with a history of seizures, neuroleptic malignant syndrome, clinically significant tardive dyskinesia, or other medical condition that would expose the subject to undue risk or interfere with study assessments.
* Subjects who are involuntarily incarcerated.
* Subjects who have undergone electroconvulsive therapy within 180 days of entry into Phase 2.
* Subjects who have used an investigational agent within 30 days of screening; and prior participation in a clinical study with aripiprazole IM depot.
* Subjects with clinically significant abnormalities in laboratory test results, vital signs, or ECG results.
* Subjects hospitalized for more than 30 days in the 90 days prior to Phase 1 (or Phase 2 for subjects bypassing Phase 1).
* Subjects requiring more than 1 benzodiazepine beyond screening (eg, lorazepam and oxazepam).
* Subjects who fail to wash-out from prohibited concomitant medications, including the use of CYP2D6 or CYP3A4 inhibitors or CYP3A4 inducers, antipsychotics, antidepressants (including monoamine oxidase inhibitors [MAOI]), and mood stabilizers, during screening and Phase 1.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 937 (Actual)
Dates: Start 2008-09; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Sanchez, MD, Study Director — Otsuka Pharmaceutical Development & Commercialization, Inc.
Locations (79):
- United States (34):
  - Cerritos, California
  - Escondido, California
  - Garden Grove, California
  - Oceanside, California
  - Orange, California
  - Pasadena, California
  - Pico Rivera, California
  - San Diego, California
  - Torrance, California
  - Washington D.C., District of Columbia
  - Gainesville, Florida
  - Kissimmee, Florida
  - Plantation, Florida
  - Tampa, Florida
  - Chicago, Illinois
  - Oak Brook, Illinois
  - Shreveport, Louisiana
  - Towson, Maryland
  - Kansas City, Missouri
  - Buffalo, New York
  - New York, New York
  - Rochester, New York
  - Hickory, North Carolina
  - South Carolina, North Carolina
  - Garfield Heights, Ohio
  - Toledo, Ohio
  - Oklahoma City, Oklahoma
  - Charleston, South Carolina
  - Johnson City, Tennessee
  - Nashville, Tennessee
  - Arlington, Texas
  - Austin, Texas
  - Richmond, Virginia
  - Milwaukee, Wisconsin
- Innsbruck, Austria
- Bruges, Belgium
- Bulgaria (6):
  - Burgas
  - Pazardzhik
  - Pleven
  - Plovdiv
  - Sofia
  - Varna
- Chile (3):
  - Santiago
  - Temuco
  - Valdivia
- Zagreb, Croatia
- Estonia (4):
  - Jämejala, Viljandimaa
  - Meegomäe
  - Tallinn
  - Tartu
- France (4):
  - Bully-les-Mines
  - Élancourt
  - Rennes
  - Saint-Nazaire
- Hungary (4):
  - Baja
  - Balassagyarmat
  - Cegléd
  - Győőor
- Italy (2):
  - Milan
  - Pisa
- Poland (9):
  - Bełchatów
  - Bialystok
  - Bydgoszcz
  - Choroszcz
  - Krakow
  - Leszno
  - Pruszków
  - Sosnowiec
  - Wroclaw
- San Juan, Puerto Rico
- South Africa (2):
  - Pretoria, Gauteng
  - Cape Town, Western Province
- South Korea (5):
  - Busan
  - Daejeon
  - Gwangju
  - Incheon
  - Seoul
- Thailand (2):
  - Muang, Chiangmai
  - Bangkok

REFERENCES:
- [Derived] Kane JM, Sanchez R, Baker RA, Eramo A, Peters-Strickland T, Perry PP, Johnson BR, Tsai LF, Carson WH, McQuade RD, Fleischhacker WW. Patient-Centered Outcomes with Aripiprazole Once-Monthly for Maintenance Treatment in Patients with Schizophrenia: Results From Two Multicenter, Randomized, Double-Blind Studies. Clin Schizophr Relat Psychoses. 2015 Summer;9(2):79-87. Epub 2015 Feb 24. PMID 25711509
- [Derived] Fleischhacker WW, Sanchez R, Perry PP, Jin N, Peters-Strickland T, Johnson BR, Baker RA, Eramo A, McQuade RD, Carson WH, Walling D, Kane JM. Aripiprazole once-monthly for treatment of schizophrenia: double-blind, randomised, non-inferiority study. Br J Psychiatry. 2014 Aug;205(2):135-44. doi: 10.1192/bjp.bp.113.134213. Epub 2014 Jun 12. PMID 24925984

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 3 phases in this study. In phases 1 and 2 (Conversion Phase and Oral Stabilization Phase), there was 1 reporting group. In phase 3 (Depot Maintenance Phase), there were 3 reporting groups. All Outcome Measures were assessed in the Depot Maintenance Phase of the study.
Groups:
- All Patients: During the Conversion Phase, patients were cross-titrated from other antipsychotics to oral non-generic aripiprazole monotherapy and during the Oral Stabilization Phase, patients were stabilized on an oral dose of aripiprazole ranging from 10 mg to 30 mg daily.
Period: Conversion Phase
Arm/Group | All Patients | Aripiprazole Depot 300 or 400 mg | Aripiprazole 10-30 mg Orally | Aripiprazole Depot 25 or 50 mg
Started | 709 | 0 (There were no patients in this reporting group in this phase of the study.) | 0 (There were no patients in this reporting group in this phase of the study.) | 0 (There were no patients in this reporting group in this phase of the study.)
Completed | 614 | 0 | 0 | 0
Not Completed | 95 | 0 | 0 | 0
Not completed — Lost to Follow-up | 4 | 0 | 0 | 0
Not completed — Sponsor Discontinued Trial | 8 | 0 | 0 | 0
Not completed — Met Withdrawal Criteria | 2 | 0 | 0 | 0
Not completed — Withdrawn by Investigator | 14 | 0 | 0 | 0
Not completed — Withdrew Consent | 38 | 0 | 0 | 0
Not completed — Adverse Event | 18 | 0 | 0 | 0
Not completed — Lack of Efficacy with Adverse Event | 9 | 0 | 0 | 0
Not completed — Lack of Efficacy without Adverse Event | 2 | 0 | 0 | 0
Period: Oral Stabilization Phase
Arm/Group | All Patients | Aripiprazole Depot 300 or 400 mg | Aripiprazole 10-30 mg Orally | Aripiprazole Depot 25 or 50 mg
Started | 842 (228 of the 842 patients who started this phase enrolled directly into this phase of the study.) | 0 (There were no patients in this reporting group in this phase of the study.) | 0 (There were no patients in this reporting group in this phase of the study.) | 0 (There were no patients in this reporting group in this phase of the study.)
Completed | 662 | 0 | 0 | 0
Not Completed | 180 | 0 | 0 | 0
Not completed — Lost to Follow-up | 17 | 0 | 0 | 0
Not completed — Sponsor Discontinue Trial | 19 | 0 | 0 | 0
Not completed — Met Withdrawal Criteria | 15 | 0 | 0 | 0
Not completed — Withdrawn by Investigator | 21 | 0 | 0 | 0
Not completed — Withdrew consent | 55 | 0 | 0 | 0
Not completed — Protocol Deviation | 2 | 0 | 0 | 0
Not completed — Adverse Event | 21 | 0 | 0 | 0
Not completed — Lack of Efficacy with Adverse Event | 20 | 0 | 0 | 0
Not completed — Lack of Efficacy without Adverse Event | 10 | 0 | 0 | 0
Period: Depot Maintenance Phase
Arm/Group | All Patients | Aripiprazole Depot 300 or 400 mg | Aripiprazole 10-30 mg Orally | Aripiprazole Depot 25 or 50 mg
Started | 0 (Patients were randomized into the 3 aripiprazole treatment groups in this phase of the study.) | 265 | 266 | 131
Completed | 0 | 196 | 178 | 61
Not Completed | 0 | 69 | 88 | 70
Not completed — Lost to Follow-up | 0 | 4 | 10 | 6
Not completed — Met Withdrawal Criteria | 0 | 4 | 6 | 5
Not completed — Withdrawn by Investigator | 0 | 8 | 12 | 8
Not completed — Withdrew Consent | 0 | 21 | 29 | 14
Not completed — Protocol Deviation | 0 | 2 | 3 | 1
Not completed — Adverse Event without Impending Relapse | 0 | 8 | 7 | 7
Not completed — Impending Relapse with Adverse Event | 0 | 13 | 12 | 17
Not completed — Impending Relapse without Adverse Event | 0 | 9 | 9 | 12

BASELINE CHARACTERISTICS:
Population: Baseline measures are based on the participants from the Depot Maintenance Phase.
Groups:
- Aripiprazole Depot 300 or 400 mg - Depot Maintenance Phase: Patients received aripiprazole 300 mg or 400 mg depot intramuscularly every 28 days for 38 weeks.
- Aripiprazole 10-30 mg Orally - Depot Maintenance Phase: Patients received aripiprazole 10-30 mg orally daily for 38 weeks.
- Aripiprazole Depot 25 or 50 mg - Depot Maintenance Phase: Patients received aripiprazole 25 mg or 50 mg depot intramuscularly every 28 days for 38 weeks.
- Total: Total of all reporting groups
Arm/Group | Aripiprazole Depot 300 or 400 mg - Depot Maintenance Phase | Aripiprazole 10-30 mg Orally - Depot Maintenance Phase | Aripiprazole Depot 25 or 50 mg - Depot Maintenance Phase | Total
Number analyzed (Participants) | 265 | 266 | 131 | 662
Age Continuous [Mean (Standard Deviation); unit: years] | 41.7 (10.4) | 41.2 (10.8) | 40.2 (9.6) | 40.7 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 98 | 53 | 256
  Male | 160 | 168 | 78 | 406

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Meeting Exacerbation of Psychotic Symptoms/Impending Relapse Criteria by the End of Week 26
Description: A patient had exacerbation of psychotic symptoms/impending relapse if they met any of the following 4 criteria. 1) Clinical Global Impression of Improvement score ≥ 5 and either an increase on any of the following Positive and Negative Syndrome Scale (PANSS) items (conceptual disorganization, hallucinatory behavior, suspiciousness, unusual thought content) to a score > 4 with an increase of ≥ 2 on that item since randomization or an increase on any of the same PANSS items to a score > 4 and an increase of ≥ 4 on the same combined PANSS items since randomization, 2) Hospitalization due to worsening of psychotic symptoms, 3) Clinical Global Impression of Severity of Suicide (CGI-SS) score of 4 or 5 on Part 1 and/or 6 or 7 on Part 2, or 4) Violent behavior resulting in clinically significant self-injury, injury to another person, or property damage.
Time Frame: Baseline to Week 26
Population: Intent-to-treat population: All randomized patients.
Measure: Number; unit: Percentage of patients
Arm/Group | Aripiprazole Depot 300 or 400 mg - Depot Maintenance Phase | Aripiprazole 10-30 mg Orally - Depot Maintenance Phase | Aripiprazole Depot 25 or 50 mg - Depot Maintenance Phase
Number analyzed (Participants) | 265 | 266 | 131
Percentage of patients | 7.12 (1.62) | 7.76 (1.72) | 21.80 (3.97)
Statistical Analysis 1: Comparison: Aripiprazole Depot 300 or 400 mg - Depot Maintenance Phase vs Aripiprazole 10-30 mg Orally - Depot Maintenance Phase; Sample sizes were estimated to achieve 93% power for the primary non-inferiority 2-sided comparison at 0.05 significance using large sample normal approximations for the distribution of the difference in binomial proportions. The assumed proportion of impending relapse at or before Week 26 for the oral aripiprazole 10-30 mg arm was 18% and the predefined non-inferiority margin was 11.5%. The sample size was projected to be 260 each for the IM depot 300 or 400 mg and oral 10-30 mg arms; Test type: Non-Inferiority or Equivalence — The test of non-inferiority of was performed using a 95% confidence interval (CI, 2-sided) for the difference in the estimated percentage of patients meeting exacerbation of psychotic symptoms/impending relapse criteria by the end of Week 26. Non-inferiority was considered confirmed if the upper bound of the 2-sided 95% CI was below the predefined margin, 11.5%; p = 0.7871, z-statistics; Mean Difference (Final Values) = -0.64, 95% CI 2-sided [-5.26 to 3.99] — The 95% CI of the difference in proportions of subjects with impending relapse events between aripiprazole IM depot 300 or 400 mg mg and oral aripiprazole were provided using the pooled SE with assumption of normality of the estimated difference
Statistical Analysis 2: Comparison: Aripiprazole Depot 300 or 400 mg - Depot Maintenance Phase vs Aripiprazole Depot 25 or 50 mg - Depot Maintenance Phase; For the superiority comparison (assay sensitivity analysis) of IM depot 300 or 400 mg to IM depot 25 or 50 mg, on a 2:1 randomization, sample sizes of 260 and 130, respectively, were calculated to provide about 95% power at the 0.05 significance level (2-sided). A superiority margin of 17% was assumed; Test type: Superiority or Other; p = 0.0006, z-statistics — Once non-inferiority was declared, superiority of depot 300/400 mg over depot 25/50 mg was tested by the difference between the proportion of subjects experiencing impending relapse by the end of Week 26 (2-sided 0.05 significance level z-statistic); The same method was used to compare IM depot 300 or 400 mg with IM depot 25 or 50 mg in the estimated proportion of subjects with impending relapse; Mean Difference (Final Values) = -14.68, 95% CI 2-sided [-23.09 to -6.27]

2. Secondary Outcome: Time to Exacerbation of Psychotic Symptoms/Impending Relapse
Time Frame: Baseline to the end of the study (Week 38)
Population: Intent-to-treat population: All randomized patients.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Aripiprazole Depot 300 or 400 mg - Depot Maintenance Phase | Aripiprazole 10-30 mg Orally - Depot Maintenance Phase | Aripiprazole Depot 25 or 50 mg - Depot Maintenance Phase
Number analyzed (Participants) | 265 | 266 | 131
Days | NA (NA) [NA to NA] — Due to the low (< 50%) percentage of relapses, median time to exacerbation could not be estimated. | NA (NA) [NA to NA] — Due to the low (< 50%) percentage of relapses, median time to exacerbation could not be estimated. | NA (NA) [NA to NA] — Due to the low (< 50%) percentage of relapses, median time to exacerbation could not be estimated.

3. Secondary Outcome: Percentage of Responders up to Week 38
Description: A patient was considered to be a responder if all of the following criteria were met. 1) Outpatient status, 2) PANSS total score ≤ 80, 3) Lack of specific psychotic symptoms on the PANSS as measured by a score of ≤ 4 on each of the following items (possible scores of 1 to 7 for each item): Conceptual disorganization, suspiciousness, hallucinatory behavior, unusual thought content, and 4) Clinical Global Impression of Severity of Illness (CGI-S) ≤ 4 (moderately ill) and 5) CGI-SS ≤ 2 (mildly suicidal) on Part 1 and ≤ 5 (minimally worsened) on Part 2.
Time Frame: Baseline to the end of the study (Week 38)
Population: Intent-to-treat population: All randomized patients.
Measure: Number; unit: Percentage of patients
Arm/Group | Aripiprazole Depot 300 or 400 mg - Depot Maintenance Phase | Aripiprazole 10-30 mg Orally - Depot Maintenance Phase | Aripiprazole Depot 25 or 50 mg - Depot Maintenance Phase
Number analyzed (Participants) | 264 | 263 | 129
Percentage of patients | 89.8 | 89.4 | 75.2
Statistical Analysis 1: Comparison: Aripiprazole Depot 300 or 400 mg - Depot Maintenance Phase vs Aripiprazole 10-30 mg Orally - Depot Maintenance Phase; Test type: Superiority or Other; p = 0.8750, z-statistics
Statistical Analysis 2: Comparison: Aripiprazole Depot 300 or 400 mg - Depot Maintenance Phase vs Aripiprazole Depot 25 or 50 mg - Depot Maintenance Phase; Test type: Superiority or Other; p = 0.0001, z-statistics

4. Secondary Outcome: Percentage of Patients Achieving Remission
Description: A patient was considered to have achieved remission if they had a score of ≤ 3 on each of the following PANSS items, maintained for a period of 6 months: Delusions (P1), unusual thought content (G9), hallucinatory behavior (P3), conceptual disorganization (P2), mannerisms/posturing (G5), blunted affect (N1), social withdrawal (N4), and lack of spontaneity (N6).
Time Frame: Baseline to the end of the study (Week 38)
Population: Intent-to-treat population: All randomized patients.
Measure: Number; unit: Percentage of patients
Arm/Group | Aripiprazole Depot 300 or 400 mg - Depot Maintenance Phase | Aripiprazole 10-30 mg Orally - Depot Maintenance Phase | Aripiprazole Depot 25 or 50 mg - Depot Maintenance Phase
Number analyzed (Participants) | 215 | 201 | 72
Percentage of patients | 48.8 | 53.2 | 59.7
Statistical Analysis 1: Comparison: Aripiprazole Depot 300 or 400 mg - Depot Maintenance Phase vs Aripiprazole 10-30 mg Orally - Depot Maintenance Phase; Test type: Superiority or Other; p = 0.3700, z-statistics
Statistical Analysis 2: Comparison: Aripiprazole Depot 300 or 400 mg - Depot Maintenance Phase vs Aripiprazole Depot 25 or 50 mg - Depot Maintenance Phase; Test type: Superiority or Other; p = 0.1097, z-statistics

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the time of the signing of informed consent until the end of the study.
Description: Safety population: All randomized subjects who received at least 1 dose of study medication.
Groups:
- All Patients - Conversion Phase: During the Conversion Phase, patients were cross-titrated from other antipsychotics to oral non-generic aripiprazole monotherapy.
- All Patients - Oral Stabilization Phase: During the Oral Stabilization Phase, patients were stabilized on an oral dose of aripiprazole ranging from 10 mg to 30 mg daily.
Arm/Group | All Patients - Conversion Phase | All Patients - Oral Stabilization Phase | Aripiprazole Depot 300 or 400 mg - Depot Maintenance Phase | Aripiprazole 10-30 mg Orally - Depot Maintenance Phase | Aripiprazole Depot 25 or 50 mg - Depot Maintenance Phase
Serious Adverse Events (participants affected / at risk) | 21/709 | 39/842 | 15/265 | 15/266 | 11/131
Other Adverse Events (participants affected / at risk) | 140/709 | 177/842 | 161/265 | 142/266 | 74/131
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients - Conversion Phase (N=709) | All Patients - Oral Stabilization Phase (N=842) | Aripiprazole Depot 300 or 400 mg - Depot Maintenance Phase (N=265) | Aripiprazole 10-30 mg Orally - Depot Maintenance Phase (N=266) | Aripiprazole Depot 25 or 50 mg - Depot Maintenance Phase (N=131)
Sick sinus syndrome (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
Drug toxicity (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Aggression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0
Hallucination, auditory (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 8 | 15 | 4 | 2 | 4
Schizoaffective disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Schizophrenia (Psychiatric disorders) | 3 | 9 | 5 | 2 | 3
Schizophrenia, paranoid type (Psychiatric disorders) | 0 | 1 | 0 | 2 | 0
Suicidal ideation (Psychiatric disorders) | 2 | 4 | 1 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Appendicitis perforated (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Ovarian fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Neuroleptic malignant syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Completed suicide (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Drug abuse (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 2 | 0 | 1 | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Aspiration pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Hernia (General disorders) | 1 | 0 | 0 | 0 | 0
Psychotic behaviour (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Transient ischemic attack (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients - Conversion Phase (N=709) | All Patients - Oral Stabilization Phase (N=842) | Aripiprazole Depot 300 or 400 mg - Depot Maintenance Phase (N=265) | Aripiprazole 10-30 mg Orally - Depot Maintenance Phase (N=266) | Aripiprazole Depot 25 or 50 mg - Depot Maintenance Phase (N=131)
Anxiety (Psychiatric disorders) | 28 | 35 | 19 | 13 | 10
Schizophrenia (Psychiatric disorders) | 5 | 7 | 3 | 3 | 8
Akathisia (Nervous system disorders) | 36 | 63 | 28 | 18 | 11
Headache (Nervous system disorders) | 39 | 44 | 26 | 30 | 7
Insomnia (Psychiatric disorders) | 78 | 87 | 31 | 37 | 18
Injection site pain (General disorders) | 0 | 1 | 20 | 6 | 1
Influenza (Infections and infestations) | 9 | 10 | 11 | 11 | 7
Nasopharyngitis (Infections and infestations) | 17 | 18 | 21 | 25 | 9
Upper respiratory tract infection (Infections and infestations) | 14 | 12 | 18 | 11 | 5
Weight decreased (Investigations) | 10 | 25 | 26 | 16 | 12
Weight increased (Investigations) | 5 | 23 | 24 | 35 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 14 | 10 | 14 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No